CLINICAL TRIAL: NCT05214846
Title: The Effect of Education and Counseling on Reducing Anxiety and Depression in Nullipar Pregnancy Women
Brief Title: Nulliparous Women and Education and Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Lecturer Dr., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/737
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy
Keywords: nulliparous momen
MeSH Terms: interventions — Educational Status; Counseling

STUDY DESIGN:
Intervention Model Description: This randomized controlled study was conducted at state hospital of nothern Turkey Obstetrics and Gynecology polyclinic between January 2021 and January 2022. The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomised controlled trials (RCTs) has been used to describe the methods.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Counseling (Experimental): After obtaining written informed consent, the data collection form, Hospital Anxiety Depression Scale (HADS) was applied to both groups by face to face interview. Immediately after the questionnaires were applied, the nurse gave individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. Women were counseled for 6 weeks.
  Anxiety-depression levels (post-test) were applied by phone call 6 weeks later.This education consisted of the definition and the purpose of pregnancy and pregnancy problems and nutrition during pregnancy, sexuality during pregnancy, number of fetal movements, preparation of the delivery bag, breast care, etc.
  Interventions: Behavioral: Education and counseling
- control group (No Intervention): Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (education and counseling) was performed.The control group was called by phone at the end of 6 weeks and told that they would be retested and 6 weeks later, they were called by phone and their anxiety and depression levels (posttest) were applied. directed to continue

INTERVENTIONS:
Behavioral: Education and counseling — After obtaining informed consent, the data collection form, Hospital Anxiety Depression Scale (HADS) was applied to both groups by face to face interview. Immediately after the questionnaires were answered, individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. In addition, the education and counseling given to the participants by the researcher.The experimental group was given a telephone number where they could receive consultancy services for 12 hours a day. Pre-test was applied. One day later, the pregnant woman was called and encouraged to call for all her questions, and she was informed that she would be returned when she called.
  Arms: Education and Counseling

SUMMARY:
This study investigates the effect of education and counseling on anxiety and depression in nullipar women.

DETAILED DESCRIPTION:
Pregnancy is a special process in a woman's life in which physiological, social and psychological changes occur. In this process, most women experience anxiety and depression, which are an important global health problem.The fear of uncertainty experienced by women who will become mothers for the first time may cause them to experience more anxiety/depression. The aim of this study was to investigate the effect of education and counseling on anxiety and depression of women.

This randomized controlled study was conducted at state hospital in northern Turkey , Obstetrics and Gynecology polyclinic between January 2022 and March 2022. Volunteer women undergoing polyclinic have been included. Participants were randomly assigned to the intervention or the control group using a computer-generated list. A data collection form including socio-demographic and obstetric characteristics such as age, educational status, Hospital Anxiety Depression Scale (HADS) was used for each patient. After obtaining written informed consent, the data collection form, Hospital Anxiety Depression Scale (HADS) were applied to both groups by face to face interview. Immediately after the questionnaires were applied, the nurse gave individual education and counseling were giving by the nurse researcher to intervention group for 30 minutes. Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (education and counseling) was performed.The IBM SPSS (Statistical package for the Social Sciences) 23.0 package program was used to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* A healthy pregnant woman over 18 years of age,
* without a diagnosed psychiatric disease,
* without mental disability and communication problems,
* at 28 weeks of gestation,
* nulliparous,
* without fetal anomaly,
* without risky pregnancy

Exclusion Criteria:

* A healthy pregnant woman under 18 years of age,
* with a diagnosed psychiatric disease,
* with mental disability and communication problems,
* under 28 weeks of gestation,
* multiparous,
* with fetal anomaly,
* with risky pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety Depression Scale (HADS) | 30 minutes
  The HADS contains 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represents 'borderline' and 0-7 'normal' (Zigmont ve Snaith).

CONTACTS AND LOCATIONS:
Overall Officials: Emine KOÇ, Asst.Prof, Principal Investigator — Ondokuz Mayıs University; Nazlı BALTACI, Asst.Prof, Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma X, Wang Y, Hu H, Tao XG, Zhang Y, Shi H. The impact of resilience on prenatal anxiety and depression among pregnant women in Shanghai. J Affect Disord. 2019 May 1;250:57-64. doi: 10.1016/j.jad.2019.02.058. Epub 2019 Feb 26. PMID 30831542
- [Background] Gonzalez-Mesa E, Kabukcuoglu K, Korukcu O, Blasco M, Ibrahim N, Cazorla-Granados O, Kavas T. Correlates for state and trait anxiety in a multicultural sample of Turkish and Spanish women at first trimester of pregnancy. J Affect Disord. 2019 Apr 15;249:1-7. doi: 10.1016/j.jad.2019.01.036. Epub 2019 Jan 31. PMID 30739036